CLINICAL TRIAL: NCT05192798
Title: A Prospective, Randomized, Open Label Clinical Study Evaluating Efficacy and Safety of Albumin-Bound Paclitaxel Combined With Antiangiogenic Agents in First-line Treatment of Relapsed or Metastatic Triple Negative Breast Cancer
Brief Title: Albumin-Bound Paclitaxel Combined With Antiangiogenic Agents in First-line Treatment of Relapsed or Metastatic TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Yan Yang, MD, Ph.D, Associate Director of the Department of Medical Oncology, The First Affiliated Hospital of Bengbu Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BYEC20211201
Record Dates: First submitted 2021-12-11; First posted 2022-01-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Triple-negative Breast Cancer
Keywords: Triple-negative breast cancer; Albumin-bound paclitaxel; Bevacizumab; Apatinib; First-line therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; apatinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group of albumin-bound paclitaxel (Active Comparator): Albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks).
  Interventions: Drug: Albumin-Bound Paclitaxel
- Group of albumin-bound paclitaxel combined with apatinib (Experimental): Albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks)+ apatinib mesylate tablet (500 mg, orally, once daily, every 3 weeks).
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Apatinib Mesylate
- Group of albumin-bound paclitaxel combined with bevacizumab (Experimental): Albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks) + bevacizumab (7.5mg/kg, intravenous infusion, once every 3 weeks).
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel — Albumin-bound paclitaxel is one of the standard first-line regimens for relapsed or metastatic triple-negative breast cancer.
Drug: Apatinib Mesylate — Apatinib mesylate is an orally administered small-molecule vascular endothelial growth factor receptor-2 (VEGFR-2) tyrosine kinase inhibitor (TKI).
  Arms: Group of albumin-bound paclitaxel combined with apatinib
Drug: Bevacizumab — Bevacizumab is a humanized anti-VEGF monoclonal antibody once approved by FDA for treatment of metastatic breast cancer in combination with chemotherapy.
  Arms: Group of albumin-bound paclitaxel combined with bevacizumab

SUMMARY:
This is a prospective, randomized, open-label clinical study. 128 patients with relapsed or metastatic triple-negative breast cancer (TNBC) who had not been systematically treated are going to be enrolled and randomly assigned to 3 groups. Group A: albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks). Group B: albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks)+ apatinib mesylate tablet (500 mg, orally, once daily, every 3 weeks). Group C: albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks) + bevacizumab (7.5mg/kg, intravenous infusion, once every 3 weeks). The dosages of therapeutic drugs are allowed to be adjusted appropriately according to the toxic reaction of the patients. Patients in three groups continued to take medication until disease progression/death/toxicity was intolerable/the patient or investigator decided to discontinue the medication.

The primary endpoint is progression-free survival (PFS). Secondary endpoints are objective response rate (ORR), clinical benefit rate (CBR, complete response (CR)+ partial response (PR) + stable disease (SD, > 6 months)), overall survival (OS), adverse events (AE), and potential predictive biomarker parameters related to treatment response (VEGF-A expression level) in peripheral blood.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is a special type of breast cancer (BC), which cannot benefit from endocrine therapy and anti-human epidermal growth factor receptor-2 (HER-2) therapy due to lack of corresponding targets. Thus, it confers a hot spot and difficulty in clinical and basic research of BC. At present, the clinical treatment of TNBC is mainly relayed on chemotherapy based on anthracycline and taxane drugs with an unsatisfactory therapeutic effects and outcomes of the patients. Although data have suggested that antiangiogenic agents may have some benefit to TNBC patients, there seems to be a lack of clinical trials evaluating efficacy and safety of albumin paclitaxel combined with antiangiogenic agents in first-line treatment of relapsed or metastatic TNBC.

This is a prospective, randomized, open-label clinical study. 128 patients with relapsed or metastatic triple-negative breast cancer (TNBC) who had not been systematically treated are going to be enrolled and randomly assigned to 3 groups. Group A: albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks). Group B: albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks)+ apatinib mesylate tablet (500 mg, orally, once daily, every 3 weeks). Group C: albumin-bound paclitaxel (260mg/m2, intravenous infusion, once every 3 weeks) + bevacizumab (7.5mg/kg, intravenous infusion, once every 3 weeks). The dosages of therapeutic drugs are allowed to be reduced, among which the lowest allowable dosage of apatinib and bevacizumab can be reduced to 250mg and 5mg/kg, respectively. The dosage of albumin-bound paclitaxel can be adjusted appropriately according to the toxic reaction of the patients. The lowest allowable dosage of albumin-bound paclitaxel can be reduced to 180mg/m2, specifically. Patients in three groups continued to take medication until disease progression/death/toxicity was intolerable/the patient or investigator decided to discontinue the medication.

The primary endpoint is progression-free survival (PFS). Secondary endpoints are objective response rate (ORR), CBR (CR+PR+SD (> 6 months)), overall survival (OS), adverse events (AE), and potential predictive biomarker parameters related to treatment response (VEGF-A expression level) in peripheral blood.

For statistical description, Kaplan-Meier method is used to plot the progression-free survival curve and estimate the median progression-free survival and its 95% confidence interval. The secondary analysis is to plot the overall survival curve using Kaplan-Meier method and estimate its 95% confidence interval. Log-rank test is used to analyze the overall survival of the main stratified factors. Objective response rate, disease control rate and 95% confidence interval are also calculated.

The safety analyses will be mainly descriptive statistical analyses, listing the incidence, severity, association, risk, and outcome of adverse events that will occur in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years and ≤80 years;
2. Patients with recurrent or metastatic triple negative breast cancer confirmed by histopathology and imaging;
3. Presence of at least one measurable lesion according to RECIST 1.1;
4. Expected survival ≥3 months;
5. Eastern Cooperative Oncology Group performance status (ECOG PS) : 0-2;
6. Patients who have not previously received antitumor systemic therapy for the stage of relapse or metastasis;
7. For subjects who have previously undergone adjuvant/neoadjuvant therapy, the time from the end of the last chemotherapy (including taxanes) to randomization should be ≥12 months; The time from the end of radical radiotherapy to randomization should be ≥6 months.
8. Major organs show good function, and the relevant examination indexes within 7 days prior to randomization meet the following requirements:

   * Absolute neutrophil count ≥ 1.5 x 10^9 / L;
   * Platelet count ≥ 100 x 10^9 / L;
   * Hemoglobin ≥ 90 g/L;
   * Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤2.5 × upper limit of normal (ULN); ALT and AST≤5 × ULN if liver metastasis is present;
   * Creatinine clearance rate(Ccr) ≥60 mL/min according to the Cockcroft-Gault formula;
   * Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5 × ULN, and international normalized ratio (INR)≤1.5 × ULN.
9. Subjects voluntarily agree to participate in the study and sign informed consent, with good compliance and being accessible for treatment and follow-up.

Exclusion Criteria:

1. Patients who are pregnant or breast-feeding;
2. Patients with multiple factors affecting oral medication (such as swallow inability, chronic diarrhea and intestinal obstruction);
3. Known hypersensitivity reaction to any of the components of the treatment;
4. Peripheral neuropathy ≥ grade 2, whatever the cause;
5. Serious other diseases as infections (hepatitis B, C and HIV), recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias or on screening, any of the following cardiac parameters: bradycardia (heart rate <50 at rest) or heart rate-corrected QT interval via Fridericia (QTcF) ≥470 msec.
6. Patients with urinary protein ≥++ indicated by routine urine examination, and the 24-hour urine protein level was confirmed to be > 1.0g;
7. Patients with imaging showing that the tumor has invaded important blood vessels or the investigator judges that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during the follow-up study;
8. Patients who have experienced arteriovenous or venous thrombosis events within 6 months prior to randomization, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism;
9. Any bleeding or bleeding event ≥grade 3 within 4 weeks prior to the first dose of therapy; Or the presence of unhealed wounds, fractures, gastrointestinal diseases such as gastric and duodenal active ulcers, ulcerative colitis, or active bleeding of unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the investigator;
10. Uncontrolled effusion management (pleural effusion, pericardial effusion, or ascites) which requires frequent drainage procedures;
11. Previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix;
12. Participants in clinical trials of other antitumor drugs within 4 weeks prior to randomization;
13. Other circumstances in which participation in the study would be inappropriate as determined by the investigator.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 2 Years.
  PFS is defined as the time from randomization until objective tumor progression or death.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | 2 Years.
  CBR is defined as the proportion of patients who have a complete, partial response or stable disease for more than 6 months to therapy.
objective response rate (ORR) | 2 Years.
  ORR is defined as the proportion of patients who have a partial or complete response to therapy.
Overall Survival (OS) | 2 Years.
  OS is defined as the time from randomization to the time of death from any cause.
Adverse Event (AE) | 2 Years.
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Serum VEGF-A | 2 Years.
  Potential predictive biomarker parameter in peripheral blood related to tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yang, M.D.,Ph.D, Principal Investigator — First Affiliated Hospital of Bengbu Medical College
Locations (1):
- Department of Medical Oncology, First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No